CLINICAL TRIAL: NCT01650896
Title: Prospective Randomised Controlled Trial of Delirium Management The Central Coast Australia Delirium Intervention Study (CADIS
Brief Title: Prospective Randomised Controlled Trial of Delirium Management by Geriatric Medicine Versus General Medicine
Acronym: CADIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Coast Local Health District (Other)
Responsible Party: Principal Investigator, Paul Regal MD FRACP FRCP (London), Senior Lecturer in Geriatric Medicine, Central Coast Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADIS-2012
Record Dates: First submitted 2012-07-10; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Delirium
Keywords: Delirium; Dementia; Instrumental activities of daily living
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General Medicine (No Intervention)
- Geriatric Medicine (Active Comparator): Daily medical review, adjust medications, treat infection, occupational therapy
  Interventions: Other: Geriatric assessment review

INTERVENTIONS:
Other: Geriatric assessment review — Adjust medications, treat precipitants of delirium, one-on-one supervision of agitated violent patients
  Arms: Geriatric Medicine

SUMMARY:
The typical delirium study between 1989 and 2005 compared delirium management in a specialty unit such as geriatric medicine with delirium management in general medicine (in most cases the research diagnosis of delirium was not communicated to the general medicine group). This study will provide open diagnosis of delirium by the CAM to both the geriatric medicine and general medicine groups (medical staff, patients, families) plus daily monitoring of delirium using digit span and delirium index which is reported to both patient groups. It will also compare confusion assessment method (CAM)to a novel diagnostic system of Paul Regal with respect to hard endpoints (survival and return home). Hypotheses: 1) General medicine can manage delirium as well as geriatric medicine when delirium is openly diagnosed and monitored daily (even in speciality units it is rare to find daily measurement of tools such as delirium index); 2) The Regal diagnostic system will be superior to the CAM in predicting hard endpoints (survival and return home rate for patients living in the community).

DETAILED DESCRIPTION:
Delirium research has been stuck in 1990 with the CAM. Articles appearing in 2012 could have been written in 1990. The CAM is riddled with logical fallacies such as 1) Circular reasoning about hearing loss causing delirium - hearing loss causes incorrect answers to questions on orientation and attention, leading to false positive diagnosis of delirium; 2) Circular reasoning on dementia causing delirium - dementia often does cause delirium but behavioral and psychological symptoms of delirium (BPSD) are the most common false positive diagnosis of delirium. CADIS (Central Coast Australia Delirium Intervention Study) will compare CAM+ to CAM- age 65+ in emergency department (prevalent delirium). Paul Regal has already shown that the 8% of 630 elderly he admitted from January 2011 to June 2012 who were CAM+ had the same survival (hospital, 90 day, 180 day and 12 month) and return home rate (65%) as 580 CAM negative elderly. The Regal criteria for delirium are completely novel. For every error in questions, the Regal system forces the examiner to determine if the error is due to poor hearing or cognitive impairment. A portable amplifier with headphones is used. The Regal methods uses recent records as the baseline for attention, memory and orientation questions. For example, an 83 year-old woman was assessed in memory clinic and had digit span forward 5/5 and 5/6; 5-word recall at 5 minutes in MoCA was 4/5; orientation was 10/10. Two months later she is admitted for RLL pneumonia and confusion. Digit span declined by 40% to 3/5, 5-word recall at 5 minutes declined by 100% to 0/5 and orientation declined by 40% to 6/10. There was no event during the two months such as stroke to explain this decline.

Another novel feature of CADIS is follow-up by a blinded clinical nurse consultant at 30 and 90 days, 12 and 24 months for MoCA, Addenbrooke Cognitve Assessment and four tests from CANTABeclipse (Cambridge Cognition) touchscreen laptop. The hypothesis is that "persistent delirium" is due primarily to irreverible brain events such as ischemic stroke.

ELIGIBILITY:
Inclusion Criteria: age 65+ medical admissions from emergency department with CAM positive delirium who have an informant / caregiver -

Exclusion Criteria: 1)Aphasia; 2) Unable to speak English; 3) End stage dementia; 4) Terminal care; 5) No close informant; 6) Unable to hear questions with or without portable amplifier with headphones; 7) Intensive care; 8) Surgical admissions

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Return home rate | 10-50 days
  The percentage of subjects returning home divided by the number living at home prior to admission and surviving until discharge
Survival | 30, 90, 180 days, 12 and 24 month
  Surivors divided by subjects reaching that milestone
Percentage residing at home | 30, 90 and 180 days, 12 and 24 months
  Number of subjects at home divided by number surviving to that milesone
Hospital complications of delirium | 7-50 days from admission
  Absconding from ward, physical violence, pulling out intravenous lines and indwelling catheters, refusing medications, falls and injurious falls

CONTACTS AND LOCATIONS:
Locations (1):
- Wyong Hospital, Kanwal, New South Wales, Australia